## **Statistical Analysis Plan**

Title

Comparative Analysis of Different Physiotherapy Interventions on Anterior Pelvic Tilt in Subjects with Non-Specific Low Back Pain: A Randomized Controlled Trial

## **DATA ANALYSIS:**

- Statistical analyses will be performed on SPSS-25.0 using appropriate methods, such as analysis of variance (ANOVA) or parametric tests (i.e paired t-test), to compare the treatment groups and determine significant differences in outcomes.
- Correlation analysis will also be done for exploring relationship between variables.
- Subgroup analyses based on demographic characteristics, pain severity, and baseline postural and balance impairments will be conducted to explore potential moderating factors.
- Test-retest reliability of the craniovertebral angle measurement will be assessed using repeated procedures and calculating ICC. Kolmogorov's test will be applied to check normality of data.

•